CLINICAL TRIAL: NCT04839185
Title: Detection of Placental Lesions in Fetal Growth Restriction
Brief Title: Placental Lesions in Fetal Growth Restrictions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1432; A532860 (Other: UW, Madison); SMPH/OBSTET & GYNECOL (Other: UW, Madison); 1U01HD087216-01 (NIH); Protocol ver: 04-06-2020 (Other: HS-IRB, UW Madison)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-05

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic: Ferumoxytol MRI (Other): The participant will receive an infusion of an iron supplement, ferumoxytol, followed by a same day MRI scan and then a second MRI scan 3-5 days later.
  Interventions: Drug: Ferumoxytol infusion; Procedure: MRI scan

INTERVENTIONS:
Drug: Ferumoxytol infusion — Ferumoxytol will be administered intravenously, by infusion, over 30 minutes. It will be used a contrast agent for MRI imaging to detect placental lesions in fetal growth restriction.
  Dose will be 255 mg in 50 mL of 0.9% Sodium Chloride Injection, USP or 5% Dextrose Injection, USP. Ferumoxytol/Feraheme will be administered only once, in one infusion of 255 mg to each subject.
  Other Names: Feraheme
Procedure: MRI scan — The MRI scanning procedure will last for approximately 60 minutes.

SUMMARY:
The purpose of this research study is to develop imaging methods to diagnose placental injury in pregnancies diagnosed with fetal growth restriction (FGR). Investigators are doing this research because the use of IV iron, followed by a Magnetic resonance imaging (MRI), may help detect injury in the placenta. The IV iron, ferumoxytol, is an iron preparation used for treatment of iron deficiency anemia. It is given in hospital setting under close medical attention. Ferumoxytol(FE) is FDA approved for some uses, but in pregnant women, its use as a MRI contrast is investigational.

DETAILED DESCRIPTION:
Research Procedure Descriptions

Blood/urine collection for research Blood and urine samples are collected at the consenting visit and at the time of delivery. A total of 10 mL, of blood is collected via venipuncture along with an aliquot of a urine sample. For research visits that coincide with clinical visits, research blood samples are collected in conjunction with clinical samples, saving subjects an additional needle stick. All subjects are asked if they wish to have left over research samples banked for future unspecified research. Blood and urine samples will be analyzed to monitor relevant maternal growth factors, multiplex assays for Cytokine panel and Matrix metalloproteinases (MMPs). Urine will be tested for Shed VE-Cadherin (VE Cad).

60 minute MRI: This MRI scan will take approximately 60 minutes. Prior to entering the MR suite, subjects are screened again for MRI safety and compatibility. The MR imaging exam is expected to take approximately 60 minutes with some additional time to get subjects comfortably placed in the scanner. Subjects are made as comfortable as possible in the bore and are provided with an alarm, which allows them to get the attention of the MR technologist conducting the scan. There is a break between scans to ensure the comfort of the subjects.

Ferumoxytol administration:

The MRI imaging with ferumoxytol as a contrast agent will be conducted at the scheduled visits based on timing of FGR diagnosis. Ferumoxytol will be administered in a hospital triage setting with maternal pulse and blood pressure monitoring and fetal heart rate monitoring. The pharmacy will be notified in advance of the arrival of the participant, so that they can prepare the infusion in a timely fashion and deliver it to triage upon participant's arrival. Participants will arrive at UnityPoint-Health Meriter Hospital obstetric triage unit as prescheduled for ferumoxytol infusion. Later that same day, the participants will present to the University of Wisconsin (UW) Hospital, Wisconsin Institutes for Medical Research (WIMR) or 1 S. Park location for their pre-scheduled MRI. In the triage unit, the nurse will obtain baseline vital signs, including maternal pulse, blood pressure, and fetal heart rate. Following this, the nurse will initiate an infusion dose of ferumoxytol. Ferumoxytol will be administered intravenously, by infusion, over 30 minutes. The participants will be monitored at 5 to 15-minute intervals, for pulse, blood pressure, respiration, and fetal heart rate. The MRI scanning procedure will be conducted at the UW Hospital, WIMR or 1 S. Park location for approximately 60 minutes.

The recommended dose of Feraheme is an initial 510 mg dose followed by a second 510 mg dose 3 to 8 days later. Investigators plan to dilute half of the recommended initial dose, i.e. 255 mg in 50 mL of 0.9% Sodium Chloride Injection, USP or 5% Dextrose Injection, USP. Feraheme will be given only once, in one infusion of 255 mg to each participant who has consented for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregravid Body Mass Index (BMI) 18.5-39.9 kg/M2
* Women with singleton pregnancies
* Ultrasound confirmed pregnancy dating prior to 14 weeks gestation
* Gestational age of 27 0/7 - 32 6/7 weeks at FGR diagnosis based on standard clinical criteria: Either estimated fetal weight (EFW) less than 10 percentile OR abdominal circumference less than 10th percentile

Exclusion Criteria:

* Diagnosis of preeclampsia at FGR diagnosis
* Gestational Diabetes Mellitus or type I/II Diabetes Mellitus
* Known fetal chromosome abnormality, structural malformation or syndromes in current pregnancy
* Known fetal viral infection syndrome
* Alcohol/drug use in current pregnancy
* History of sickle cell anemia, sickle cell trait or other inherited anemia with risk of iron overload
* Contraindications to MRI (such as claustrophobia, metallic implant, etc.) based on MRI Screening
* Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Any physical or psychological symptom, based on the clinical judgment of the study physician that would make a participant unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Shah, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from UnityPoint Health-Meriter Hospital, April 2021 to July 2021.
Groups:
- Diagnostic: Ferumoxytol MRI: The participant will receive an infusion of an iron supplement, ferumoxytol, followed by a same day MRI scan and then a second MRI scan 3-5 days later.
  Ferumoxytol infusion: Ferumoxytol will be administered intravenously, by infusion, over 30 minutes. It will be used a contrast agent for MRI imaging to detect placental lesions in fetal growth restriction.
  Dose will be 255 mg in 50 mL of 0.9% Sodium Chloride Injection, USP or 5% Dextrose Injection, USP. Ferumoxytol/Feraheme will be administered only once, in one infusion of 255 mg to each subject.
  MRI scan: The MRI scanning procedure will last for approximately 60 minutes.
Period: Overall Study
Arm/Group | Diagnostic: Ferumoxytol MRI
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic: Ferumoxytol MRI
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2
  40-49 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which Intervillous Placental Blood is Detected
Description: Intervillous Placental Blood will be detected by Magnetic resonance imaging (MRI). The patient will receive the first 60-minute MRI within 1-15 hours after completion of the ferumoxytol infusion.
Time Frame: up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic: Ferumoxytol MRI
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Number of Participant for Which Placental Lesions Are Detected
Description: Placental lesion will be detected by Magnetic resonance imaging (MRI). The patient will receive the first 60-minute MRI within 1-15 hours after completion of the ferumoxytol infusion.
Time Frame: up to 1 week
Population: Please see Limitations and Caveats section
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic: Ferumoxytol MRI
Number analyzed (Participants) | 3
Participants | 2

3. Primary Outcome: Number of Participants for Which Macrophage at the Implementation Site Are Detected
Description: FE-MRI (ferumoxytol- magnetic resonance imaging) will be used first time as a contrast agent to generate for the 3D high-resolution MRI maps of macrophages at the maternal-fetal interface (MFI) in real time in vivo.
Time Frame: up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic: Ferumoxytol MRI
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events data will be collected from when the participant signs consent through 6 week post-partum, or up to 3 months on study.
Arm/Group | Diagnostic: Ferumoxytol MRI
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic: Ferumoxytol MRI (N=3)
Headache (Nervous system disorders) | 1
Abdominal Cramp (Gastrointestinal disorders) | 1
Upper Respiratory Viral Infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
There is not enough data to conclusively categorize placental lesions due to a lack of comparative normative placental data or targeted biopsy, which would require advanced novel methodology to match locations in imaging data with pathology data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT04839185/Prot_SAP_000.pdf